CLINICAL TRIAL: NCT00153439
Title: Purdue University Parenting Program Attrition and Compliance Efficacy Trial
Brief Title: Purdue University Parenting Program Attrition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Purdue University (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: CDC-NCIPC-3928; R49/CCR522339-03
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2007-09-10 (Estimated); Status verified 2007-09

CONDITIONS: Child Abuse
Keywords: parenting; motivation; child maltreatment; program attrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Motivational enhancements, parent training

SUMMARY:
The purpose of this study is to examine the efficacy of techniques to enhance participation in parenting programs.

DETAILED DESCRIPTION:
This project addresses the problem of involving parents in interventions that promote parenting effectiveness and child coping-competence in preschoolers as a means of reducing risk of child maltreatment (and related adverse developmental outcomes). Purdue University will examine the impact of partnership (organizational involvement in recruitment and retention), cash incentives, and a motivational goal setting component on participation and engagement in the Parenting Our Children to Excellence program, a group intervention for parents and caregivers of preschool children.

ELIGIBILITY:
Inclusion Criteria:

* Parents with children 3-5 years old who attend centers in which interventions are offered

Exclusion Criteria:

* See above. No other exclusion criteria will be used.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 560
Dates: Start 2003-07; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Engagement and participation in an 8-week parenting program

SECONDARY OUTCOMES:
Measures of parenting behavior and attitudes, incidents of child maltreatment, measures of child adjustment and functioning

CONTACTS AND LOCATIONS:
Overall Officials: Jean E Dumas, Ph.D., Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States